CLINICAL TRIAL: NCT02481934
Title: Phase 1 Clinical Trial to Evaluate Security and Dose of Expanded and Activated Autologous NK Cells Infusions in Consolidation of Multiple Myeloma Patients Treatment on Second or Later Relapse.
Brief Title: Clinical Trial of Expanded and Activated Autologous NK Cells to Treat Multiple Myeloma
Acronym: NK-VS-MM
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Joaquín Martínez López, MD, PhD (Other)
Collaborators: Hospital Infantil Universitario Niño Jesús, Madrid, Spain (Other)
Responsible Party: Sponsor-Investigator, Joaquín Martínez López, MD, PhD, Hematology Head of department, M.D., Ph.D., Hospital Universitario 12 de Octubre
Organization: Hospital Universitario 12 de Octubre (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NK-VS-MM
Record Dates: First submitted 2015-06-10; First posted 2015-06-25 (Estimated); Results first posted 2016-12-05 (Estimated); Last update posted 2021-08-20 (Actual); Status verified 2021-08

CONDITIONS: Multiple Myeloma
Keywords: Recurrent multiple myeloma; NK cells; cell therapy; NKAE; Relapsed multiple myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Lenalidomide; Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NKAE cells infusion + chemotherapy (Experimental): Expanded and activated autologous NK cells (NKAEs) + chemotherapy (lenalidomide OR bortezomib).
  Interventions: Procedure: NKAE cells infusion; Drug: Lenalidomide; Drug: Bortezomib

INTERVENTIONS:
Procedure: NKAE cells infusion — Expanded and activated autologous NK cells infusion. Each patient will receive two infusions of 7.5 x 106 expanded and activated autologous NK cells/kg/cycle.
  Other Names: NKAE infusion; Activated and expanded autologous NK cells infusion
Drug: Lenalidomide — Lenalidomide, 10 mg oral/day during 21 days (cycle). Patients will receive 4 cycles.
  Other Names: Revlimid
Drug: Bortezomib — Bortezomib, 1.3 mg/m2, s.c., days 1, 4, 8 and 11/cycle. Patients will receive 4 cycles.
  Other Names: Velcade

SUMMARY:
The purpose of this study is to determine wether activated and expanded autologous Natural Killer cells (NKAEs) are effective in the treatment of patients with multiple myeloma on second or later relapse. NKAEs are used in combination with anti-myeloma drugs such as lenalidomide or bortezomib.

DETAILED DESCRIPTION:
It is expected to enroll 10 to 15 patients within 18 months. Patients have to achieve stable disease after induction therapy. Peripheral blood from patients will be collected every cycle (n=4) to produce NKAEs under Good Manufacturing Practice (GMP) conditions peripheral blood mononuclear cell (PBMCs) will be co-cultured with a genetically modified cell line (K562-mb15-41BBL) and 100 IU/ml interleukin-2.

Treatment consists of 4 cycles of anti-myeloma consolidation treatment with two infusions of NKAEs every day 1 and 8 of each cycle. Usually, chosen treatment regime will be bortezomib (Velcade) or lenalidomide (Revlimid). These treatments are used to be combined with corticosteroid medications which needs to be suspended before NKAEs infusions. A washout period of 2 weeks is required.

NKAEs dose of cells will be constant, 7.5x106/kg. There will be an interim analysis intra-cohort one week after the first batch of two infusions. If at the analysis no grade IV adverse effect is observed we will proceed to the second cycle and the inclusion of other patients.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between 20 and 80 years old
* With multiple myeloma in 2nd or later relapse or showing resistance after 2 treatment lines
* Eastern Cooperative Oncology Group (ECOG) ≤ 2
* Life expectancy greater than six months
* Creatinine clearance rate more than 30 ml / min
* Subjects who have received at least 4 cycles of rescue treatment under the procedures of the 12 de Octubre Hospital (rescue treatment will vary depending on previous anti-myeloma treatment). After treatment, patients must have shown chemosensitivity and disease stabilization.
* Will be included subjects with partial response or stable disease (for at least 2 cycles) after 75% of planned rescue treatment or patients at subclinical progression (defined as an increase of monoclonal component ≥ 25%) at any time of rescue treatment. Subjects have to show tolerance to rescue treatment, without G3/4 adverse effects, if G1/2 adverse effects exist they must be analyzed immediately before starting reinfusion program.
* Subjects have to agree to participate in the trial and they have to sign informed consent.

Exclusion Criteria:

* Subjects with clinical progression or complete response will not be included.
* Any of the following abnormal laboratory results:

Absolute Neutrophil Count < 1000/ µL Platelets Count < 50000/ µL in those patients with bone marrow infiltration lower than 50% Measured creatinine clearance <30 ml/min Hemoglobin level ≤ 8 g/dL Peripheral neuropathy ≥ Grade 2

* Subjects have received allogeneic stem cell transplant.
* Subjects with heart disease which compromises patient's life or protocol accomplishment.
* Subjects with past clinical history of malignant disease within 3 years (exceptions are squamous or basal cell carcinoma).
* Subjects receiving another investigational drug or having received investigational drug within 30 days before screening.
* Subjects who require chronic steroid or immunosuppressive treatment.
* Any condition, including abnormally laboratory results, that might compromise the patient´s life if he participate in this study.
* Any concurrent medical condition, abnormally laboratory results or any psychological disorder that prevent the patient to sign the informed consent.
* Pregnant or fertile women.
* Patients known to be seropositive for human immunodeficiency virus (VIH) or having active hepatitis A, B or C.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2013-03; Primary Completion 2016-07 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joaquín Martínez López, M.D, Ph.D, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was performed between march 2013 and october 2014 at Hospital 12 de Octubre in Madrid.
Period: Overall Study
Arm/Group | NKAE Cells Infusion + Chemotherapy
Started | 5
Completed | 3
Not Completed | 2
Not completed — Death | 2

BASELINE CHARACTERISTICS:
Population: The number of participants was directly related with the cost of expanded and activated NK cells production.
Groups:
- NKAE Cells Infusion + Chemotherapy: Expanded and activated autologous NK cells (NKAEs) + chemotherapy (lenalidomide OR bortezomib).
  NKAE cells infusion: Expanded and activated autologous NK cells infusion. Each patient will receive: two infusions of 7.5 x 106 expanded and activated autologous NK cells/kg/cycle.
  Lenalidomide: Lenalidomide, 10 mg oral/day during 21 days (cycle). Patients will receive 4 cycles.
  Bortezomib: bortezomib, 1.3 mg/m2, s.c., days 1, 4, 8 and 11/cycle. Patients will receive 4 cycles.
Arm/Group | NKAE Cells Infusion + Chemotherapy
Number analyzed (Participants) | 5
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 62 [61 to 72]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 2
Region of Enrollment [Number; unit: participants]
  Spain | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events During NKAE Treatment
Description: Toxicity will be assessed by adverse events count during NKAE treatment monitoring peripheral blood absolute neutrophil count (cells/μl). Toxicity will be evaluated monthly during NKAE treatment (4 months). During follow-up, it will be assessed monthly the first 6 months. After that, quarterly until one year of follow-up, based on Common Toxicity Criteria for Adverse Events of the National Cancer Institute (CTCAE) to v.4.03.
Time Frame: 16 months
Population: Analysis per protocol
Measure: Number; unit: participants
Arm/Group | NKAE Cells Infusion + Chemotherapy
Number analyzed (Participants) | 5
participants | 2

2. Secondary Outcome: Number of Participants With Peripheral Blood Monoclonal Protein Reduction or Stabilization
Description: Efficacy will be assessed monthly during NKAE treatment (4 months) by peripheral blood monoclonal protein monitoring. During follow-up, efficacy will be evaluated monthly the first 6 months. After that, quarterly until one year of follow-up.
Time Frame: 16 months
Measure: Number; unit: participants
Arm/Group | NKAE Cells Infusion + Chemotherapy
Number analyzed (Participants) | 5
participants | 5

ADVERSE EVENTS:
Time Frame: 4 months during treatment with NKAE cells.
Arm/Group | NKAE Cells Infusion + Chemotherapy
Serious Adverse Events (participants affected / at risk) | 2/5
Other Adverse Events (participants affected / at risk) | 2/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKAE Cells Infusion + Chemotherapy (N=5)
Gastrointestinal bleeding (Gastrointestinal disorders) | 1 (1) — The patient was suffering for gastrointestinal bleeding before enrollment.
Vertebral compression (Musculoskeletal and connective tissue disorders) | 1 (2) — This serious adverse event was due to multiple myeloma bone lesions.
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | NKAE Cells Infusion + Chemotherapy (N=5)
Neutropenia (Immune system disorders) | 2 (2) — Two patients had grade II neutropenia but none of them need dose adjustment.

LIMITATIONS AND CAVEATS:
Volume of the peripheral blood from patients was limiting in order to perform different cohorts with more NKAE cells infusions.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No